CLINICAL TRIAL: NCT01284101
Title: Prospective Randomized Study Comparing Endothelial Cell Loss Using the Tan EndoGlide With Forceps for Insertion of the Donor Graft in DSAEK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. Allan Slomovic, Toronto Western Hospital, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB-10-0632-B
Record Dates: First submitted 2011-01-24; First posted 2011-01-26 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Endothelial Cell Loss With Different Insertion Devices
MeSH Terms: interventions — Surgical Instruments

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Forceps delivery of donor graft (Active Comparator): Using the forceps to insert the donor graft.
  Interventions: Device: Forceps for delivery of the donor graft
- Tan Endoglide for insertion of the donor graft (Experimental): Use of the Tan Endoglide for insertion of the donor graft.
  Interventions: Device: Use of the Tan Endoglide to insert the donor graft

INTERVENTIONS:
Device: Use of the Tan Endoglide to insert the donor graft — Using the Tan Endoglide to insert the donor graft into the eye
  Arms: Tan Endoglide for insertion of the donor graft
Device: Forceps for delivery of the donor graft — Use of the forceps for delivery of the donor graft into the eye.
  Arms: Forceps delivery of donor graft

SUMMARY:
The Tan EndoGlide device results in less endothelial cell trauma during insertion of the donor corneal graft indicated by reduced endothelial cell loss at 1 year follow-up compared to the Forceps.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with corneal decompensation requiring DSAEK with or without cataract surgery for visual rehabilitation.
* Clinical diagnosis include endothelial cell dysfunction secondary to Fuchs endothelial dystrophy, pseudophakic or aphakic bullous keratopathy, failed penetrating keratoplasty or DSAEK, iridocorneal endothelial syndrome or trauma.
* Ability to understand the nature of the procedure and give full informed consent.
* Patients who are able to comply with the standard DSAEK follow-up protocol at the Toronto Western Hospital.

Exclusion Criteria:

* Patients with late stage corneal decompensation with stromal scarring unsuitable for DSAEK and therefore requiring penetrating keratoplasty.
* Patients with complex anterior segment pathology precluding successful DSAEK procedure.
* Patients not giving full informed consent to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Donor Graft Endothelial cell counts | 1 year
Best corrected visual acuity | 1 year

SECONDARY OUTCOMES:
Complications of surgery | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada